CLINICAL TRIAL: NCT02387775
Title: Temperature Control With an Esophageal Cooling Device: A Feasibility Study in Post Cardiac Arrest Patients
Brief Title: Temperature Control With an Esophageal Cooling Device in Post Cardiac Arrest Patients
Acronym: E-Chill
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Western University, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 106185
Record Dates: First submitted 2015-03-09; First posted 2015-03-13 (Estimated); Last update posted 2018-07-30 (Actual); Status verified 2018-05

CONDITIONS: Anoxic Brain Injury; Cardiac Arrest
Keywords: esophageal cooling device; post cardiac arrest; targetted temperature management; therapeutic hypothermia; cooling; rewarming
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Esophageal temperature control (Experimental): The Esophageal Cooling Device (ECD) will be inserted and utilized for temperature control for up to 36 hours in this arm. The ECD will be used for all three phases of therapeutic hypothermia; induction, maintenance, and rewarming. Conventional cooling or warming techniques (e.g. cold saline, ice packs, cooling or warming blankets) will still be made available to the treating ICU team to be used at their discretion.
  Interventions: Device: Esophageal temperature control

INTERVENTIONS:
Device: Esophageal temperature control — Insertion of the Esophageal Cooling Device (ECD) will take place as described in the product monograph. The ECD will be connected to the heat exchange unit Blanketrol Hyper-Hypothermia System® (Cincinnati Sub-Zero, Cincinnati, OH) and will be used for temperature control for a total of 36 hours. A patient target of 35°C will be set on the heat exchange unit. Once target is attained, it will be maintained for 24 hours. Slow rewarming will then be achieved by increasing the input target by 0.2°C per hour, until a target of 36.6°C is reached.
  All temperature data (device, input target, and patient bladder temperature) will be captured automatically using Data Export Software® (Cincinnati Sub-Zero, Cincinnati, OH) on an external laptop connected to the external heat exchange unit.
  Other Names: Esophageal Cooling Device®

SUMMARY:
This is a prospective, interventional study aiming to assess the effectiveness of the Esophageal Cooling Device (ECD) as a temperature control modality in post cardiac arrest patients. In addition, observed adverse events during ECD use, ease-of-use, nurse satisfaction and patient outcomes will be examined.

DETAILED DESCRIPTION:
Temperature control in comatose survivors of cardiac arrest, is a critical aspect of these patients' care. In this context, mild temperature reduction for 24 hours post cardiac arrest has been shown to improve neurological outcomes.

Hypothermia is commonly induced using a combination of internal and external cooling modalities. Internal cooling modalities include intravenous administration of cold crystalloids and intravascular cooling catheters. External or body surface cooling can be achieved using cooling blankets, adhesive pads, and ice packs. Each of these methods however, has its limitations.

Administration of intravenous refrigerated crystalloid (4°C) boluses is a simple, effective and widely available method of hypothermia induction. Lack of precise temperature control and the potential for pulmonary edema however, make this modality unsuitable for the maintenance phase of hypothermia. Surface cooling methods, such as cooling blankets and ice packs, often cause shivering, skin breakdown, and in obese patients may be ineffective. Intravascular cooling catheters require the time of a physician for insertion and bear the potential risks of line infection and deep venous thrombosis. Searching for a temperature control device that overcomes the limitations, inefficiencies and inconveniences of existing modalities is therefore strongly desired.

The ideal temperature control modality should be effective, predictable and easy to use. An esophageal cooling device has recently become available which in theory may, may possess some of these attributes. To date, there have been no published studies examining this device's efficacy. In addition, no study has documented any adverse events during it's use, or evaluated it's ease-of-use at the bedside.

This is a prospective, interventional study aiming to assess the effectiveness of the Esophageal Cooling Device (ECD) as a temperature control modality in comatose survivors of cardiac arrest (the E-Chill trial). In addition, observed adverse events during ECD use, ease-of-use, nurse satisfaction and patient outcomes will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the intensive care unit after resuscitation from an out-of-hospital cardiac arrest.
* Sustained return of spontaneous circulation (no chest compressions required for >20 minutes)
* Not obeying commands to verbal instruction.
* On mechanical ventilation via endotracheal tube or tracheotomy.

Exclusion Criteria:

* Known esophageal deformity (known esophageal varices, history of esophagectomy, previous swallowing disorders, achalasia, etc.) or evidence of esophageal trauma.
* Known ingestion of acidic or caustic poisons within the prior 24 hours.
* Patients with less than 40 kg of body mass.
* Patients known to be pregnant.
* Uncontrolled coagulopathy.
* Documented intracranial hemorrhage.
* Patients presenting to the intensive care unit with a temperature < 35°C.
* Time from collapse to return of spontaneous circulation > 45 minutes or unknown.
* Time from collapse to starting chest compressions > 10 minutes or unknown.
* Time from collapse to assessment for enrollment > 12 hours.
* Patients thought to have a very low chance of surviving the next 48 hours as assessed by the research team.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-12; Primary Completion 2018-06 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Percent of time maintained within 0.5°C range of the 35°C input target, in the hypothermia maintenance phase. | Within 36 hours of ECD insertion.
  Once patient temperature is within 0.5°C from the 35°C target, the maintenance phase will commence. The amount of time patient temperature is maintained within ± 0.5 from 35°C, as a percentage of the total hypothermia maintenance time (24 hours) will be examined. Confidence intervals for the results will be reported.

SECONDARY OUTCOMES:
Cooling rate in hypothermia induction phase. | Within 10 hours of ECD insertion.
  Average rate of temperature drop during the hypothermia induction phase. The induction phase ends once the patient temperature is within ± 0.5 from the 35°C target. Confidence intervals for the results will be reported.
Percent of time patient temperature is within 0.5°C range of the input target, 30 minutes after each target elevation in the rewarming phase. | Within 36 hours of ECD insertion.
  Rewarming time will be considered to start, 30 minutes after the input target is increased from 35 to 35.2°C. Since patient temperature is likely to change slowly after that change, the recorded temperature taken 30 minutes after the target change will be used. Therefore if the target temperature is changed to 35.2°C at noon, the patient temperature recorded at 12:30 will be used. Whether or not the patient is within ± 0.5 from the 35.2°C target will be calculated using the patient temperatures recorded at 12:30 till the next change in target temperature. And for each subsequent elevation in target, this same rule will be applied. This calculation will be taken to reflect the degree of control over rewarming. Confidence intervals for the results will be reported.
ECD insertion time. | Within 4 hours of enrollment.
  Time taken to insert the Esophageal Cooling Device (ECD) will be measured. This will only include time needed to insert the ECD orally and advance it to the appropriate depth. This will exclude the steps prior to insertion (measuring the appropriate depth of insertion externally, connecting the ECD to the external heat exchange unit, and lubing the tip of the ECD). Taping the ECD in place will be excluded from this time recording as well.
Adverse events during and after ECD use. | Within 4 weeks of enrollment or until hospital discharge whichever comes first.
  Recorded events during or after ECD use: cardiac arrhythmias, bradycardias, myocardial infarction/re-infarction, ventilator associated pneumonia, gastrointestinal bleeding (any), esophageal injury, dysphagia, odynophagia, aspiration pneumonia, non-aspiration pneumonia, tube feed intolerance, reflux and evidence of esophagitis.
Ease-of-use. | Within 40 hours of enrollment.
  Nurses taking care of patients with the device will be asked to rate the following:
  I. Observed ease of insertion of device 1 = poor, 3 = average, 5 = excellent. II. General ease-of-use and handling: 1 = poor, 3 = average, 5 = excellent. III. How the ECD compares to our standard methods of inducing hypothermia: 1 = inferior, 3 = equivalent, 5 = superior.
  IV. Since ECD insertion, have any other cooling modality been used to cool or warm the patient? If yes, please specify.
Patient neurological outcome as defined by the Cerebral Performance Category. | Within 4 weeks of enrollement or until hospital discharge whichever comes earlier.
  Patient neurological outcome will be dichotomized into good or bad. Good outcome will be equivalent to CPC scores of 1 & 2 (where the patient is independent), and bad outcome will be equivalent to CPC scores of 3, 4 & 5 (where the patient is either dependent or dead).
  CPC Scale:
  1. Functioning normally and independent, possibly with a minor disability.
  2. Moderately disabled, still independent.
  3. Conscious but with a severe disability, dependent.
  4. Unconscious (comatose or in a persistent vegetative state).
  5. Brain dead or dead by traditional criteria.
Need for other cooling or warming modalities during ECD use. | Within 36 hours of ECD insertion.
  The requirement for any of the following cooling modalities during ECD use will be documented.
  1. Intravenous refrigerated saline. Data collected: times of use, volumes administered, and reasons for use as per bedside nurse.
  2. Cooling or warming blanket use. Data collected: times of use, duration of application, and reason for use as per bedside nurse.
  3. Ice-pack application. Data collected: time of use, body location(s) applied, duration of application, and reason for application as per bedside nurse.
  4. Body cavity cold fluid irrigation e.g. bladder, peritoneal... etc. Data collected: time of use, body cavity site, reason for use as per bedside nurse.

OTHER OUTCOMES:
Shivering during ECD use. | Within 36 hours of ECD insertion.
  The development of shivering in patients not receiving neuromuscular blockade during ECD use will be examined. This will not be evaluated however, in patients receiving neuromuscular blockade as part of their hypothermia protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed F. Hegazy, MBBCh, FRCPC, Principal Investigator — Western Univeristy, Canada
Locations (2):
- Canada (2):
  - University Hospital, London Health Sciences Centre, University of Western Ontario, London, Ontario
  - Victoria Hospital, London Health Sciences Centre, University of Western Ontario, London, Ontario

REFERENCES:
- [Background] Hegazy AF, Lapierre DM, Butler R, Althenayan E. Temperature control in critically ill patients with a novel esophageal cooling device: a case series. BMC Anesthesiol. 2015 Oct 19;15:152. doi: 10.1186/s12871-015-0133-6. PMID 26481105
- See also: The esophageal cooling device insertion steps, the heat exchange unit set-up, our local practice at London Health Sciences Centre, and some general recommendations on the device's use. — https://www.youtube.com/watch?v=I3_tySqrwQk